CLINICAL TRIAL: NCT05846516
Title: A Phase 1b Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of a Heterologous Prime Boost Vaccination (ATP150/ATP152/ATP162, VSV-GP154) and Ezabenlimab (BI 754091) in Patients With Pancreatic Ductal Adenocarcinoma.
Brief Title: A Study to Test KISIMA-02 Vaccine-based Immunotherapy and Ezabenlimab in People With Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1515-0001
Record Dates: First submitted 2023-04-18; First posted 2023-05-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental)
  Interventions: Drug: VSV-GP154; Drug: ATP150; Drug: ATP152
- Cohort B (Experimental)
  Interventions: Drug: VSV-GP154; Drug: ATP150; Drug: ATP152; Drug: Ezabenlimab
- Cohort C Treatment (Experimental)
  Interventions: Drug: VSV-GP154; Drug: Ezabenlimab; Drug: ATP162
- Cohort C Observational (No Intervention)

INTERVENTIONS:
Drug: VSV-GP154 — VSV-GP154
  Arms: Cohort A; Cohort B; Cohort C Treatment
Drug: ATP150 — ATP150
  Arms: Cohort A; Cohort B
Drug: ATP152 — ATP152
  Arms: Cohort A; Cohort B
Drug: Ezabenlimab — Ezabenlimab
  Arms: Cohort B; Cohort C Treatment
Drug: ATP162 — ATP162
  Arms: Cohort C Treatment

SUMMARY:
This study is open to adults with advanced pancreatic cancer. The study tests a type of immunotherapy. It is a protein treatment combined with a virus that may kill cancer cells and help the immune system fight cancer. The immunotherapy is combined with a study medicine called ezabenlimab. Ezabenlimab is an antibody that may also help the immune system fight cancer.

The purpose is to find the highest dose of the immunotherapy that people with pancreatic cancer can tolerate when taken alone or together with ezabenlimab (Part A and B). To find out, researchers look at the number of participants with certain severe health problems. The purpose of Part C is to check whether the immunotherapy combined with ezabenlimab may increase survival. Participants are put randomly into 2 groups. One group receives the immunotherapy combined with ezabenlimab and the other group receives standard treatment. Researchers compare the results between the groups.

Participants can stay in the study as long as they tolerate the treatment or up to 1 year. During that time, they regularly visit the site. At all visits, the doctors closely check the health of the participants and note any severe health problems.

ELIGIBILITY:
Key inclusion criteria

* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC)
* ECOG performance status of 0 or 1.
* Patients with advanced or metastatic disease who completed at least 16 weeks of standard of care systemic chem-/chemoradiotherapy and achieved a partial response or stable disease.
* Patients who underwent confirmed R0 or R1 resection and completed at least 3 months of combined peri-adjuvant multiagent chemotherapy.
* No evidence of disease progression or recurrence.
* Start of study treatment within 12 weeks from the last curative treatment (resected PDAC).
* Patient must have completed 8-12 cycles of FOLFIRINOX or mFOLFIRINOX either as adjuvant, neoadjuvant, or perioperative (Part C)
* Life expectancy at least 12 months (resected PDAC), or at least 6 months (advanced/metastatic PDAC).
* Archival tumor tissue availability for central KRAS analysis and research.

Key exclusion criteria

* Not yet recovered from surgery (resected PDAC).
* Gastro-intestinal bowel obstruction.
* Other malignancy within the last 3 years.
* Prior chemotherapy or targeted small molecule therapy within 14 (locally advanced/metastatic PDAC) or 28 (resected PDAC) days from initiation of study treatment.
* Prior radiotherapy within 14 days (advanced/metastatic PDAC). No prior radiotherapy. in resected PDAC
* Prior use of immunotherapeutic agents, including but not limited to checkpoint inhibitors or VSV-based agents.
* Diagnosis of immunodeficiency, and/or history of allogeneic organ transplant
* Chronic systemic treatment with steroids or other immunosuppressive medications.
* Active autoimmune disease requiring systemic treatment within the last 2 years.
* Chronic or concurrent active infectious disease requiring systemic antibodies, antifungal, or antiviral treatment
* Major (according to the Investigator's judgment) surgery within 12 weeks from initiation of study treatment
* Use of Tamoxifen within 1 month prior to start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2029-02-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity (DLT) | Over at least 35 days
  Part A and B
Disease-free survival (DFS), defined as the time from randomization until confirmed relapse or death from any cause, whichever occurs earlier. | Through study completion, an average of 24 months.
  Part C

SECONDARY OUTCOMES:
Proportion of patients with clearance and normalization of tumor biomarkers | Up to 12 months
  Part B and C
Occurrence of dose-limiting toxicity (DLT) during the on-treatment period | Throughout the study, up to 12 months.
  Part B and C

CONTACTS AND LOCATIONS:
Locations (20):
- United States (12):
  - University of Southern California, Los Angeles, California
  - University of California Los Angeles, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Asklepios Kliniken Hamburg GmbH, Hamburg, Germany
- Spain (4):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Clara Campal Comprehesive Cancer Center, Madrid
- Switzerland (3):
  - University Hospital Bern, Bern
  - Hopitaux Universitaires de Geneve (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com